CLINICAL TRIAL: NCT04149080
Title: Effects on Bone Neoformation of Simvastatin Gel Covered With Polypropylene Membrane in Post-extraction Sockets: a Randomized Controlled Trial
Brief Title: Effects of Simvastatin Gel on Bone Neoformation in Post-extraction Sockets: a Randomized Controlled Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidade Federal Fluminense (Other)
Responsible Party: Principal Investigator, Rebecca Cruz, MSc., Universidade Federal Fluminense
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: SIM01
Record Dates: First submitted 2019-10-30; First posted 2019-11-04 (Actual); Last update posted 2019-11-04 (Actual); Status verified 2019-10

CONDITIONS: Alveolar Socket Preservation; Bone Regeneration
Keywords: Simvastatin; Tooth extraction; Alveolar socket preservation; Bone regeneration

STUDY DESIGN:
Intervention Model Description: 30 subjects will be divided randomly in two groups. The study is triple masked.
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SIM Group (Experimental): Alveolar socket post-extraction filled with Simvastatin covered with polypropylene membrane
  Interventions: Procedure: SIM + polypropylene membrane
- Control Group (Placebo Comparator): Alveolar socket post-extraction covered with polypropylene membrane
  Interventions: Procedure: Placebo

INTERVENTIONS:
Procedure: SIM + polypropylene membrane — After tooth extraction the socket will be filled with 1.2% simvastatin gel and covered with polypropylene membrane, which will be intentionally exposed.
  Arms: SIM Group
Procedure: Placebo — After tooth extraction the socket will be filled with gel and covered with polypropylene membrane, which will be intentionally exposed.
  Arms: Control Group

SUMMARY:
Statins (HMG-CoA) are widely used in treating patients with hypercholesterolemia. They have also been studied because of their anabolic effects on bone tissue. Statins increase the expression of Bone Morphogenetic Proteins-2 (BMP-2) and Vascular Endothelial Growth Factor (VEGF), which are of important scientific interest in bone regeneration therapy. However, they are expensive and have a short half-life. Therefore, a molecule promoting the endogenous production of BMP-2 and VEGF would be valuable for the field of bone tissue engineering. This study aims to evaluate dimensional changes, level of soft tissue healing, pain/discomfort, and newly formed tissues in post-extraction sockets filling with Simvastatin (SIM) gel covered with polypropylene membranes. Thirty post-extraction sockets of posterior teeth will be randomized allocated in two groups: 1) extractions and socket filling with 1.2% SIM gel and membrane and 2) extraction and socket filling with placebo gel and membrane. The evaluation will be done through clinical analyzes, histomorphometry and micro-computed tomographic images, considering the dimensional changes, the quantity and the quality of tissue formation after extractions. Measurements will be taken before extraction (T1) and 90 days after the extraction (T2). In addition, the perception of pain will be analyzed. The hypothesis is that SIM associated with polypropylene membrane can enhance bone formation in post-extraction sockets compared with the control group.

DETAILED DESCRIPTION:
This study will be a triple masking randomized controlled trial, being conducted according to the principles outlined in the Declaration of Helsinki regarding experiments on human subjects. This work was submitted to the Ethics Committee of Antonio Pedro University Hospital, with the approval number: 71087917.4.0000.5243. Consort checklist will be followed as a guideline to ensure the quality and transparency of this research.

The volunteers are being recruited at the Dental Clinical Research Center of the Fluminense Federal University and they have to agree to participate in the study, signing the consent form and being willing to follow the guidelines and timelines. The sample will consist of 30 human alveolar sockets, where the teeth involved should provide indication of tooth extraction without treatment possibilities after clinical and radiographic examination.

Dental and medical records of all volunteers will be checked. Furthermore, they will have a clinical examination and tomography. Before surgery, all volunteers will undergo basic periodontal therapy and oral hygiene instructions. The primary outcome variables included soft and hard tissue (measured in millimetres), assessed using customized acrylic templates and tomography, performed before surgery standardize the initial (T1) and final measurements (T2) 90 days after tooth extraction. Secondary outcomes included the level of soft tissue healing, pain/discomfort reported by the participants, and representative histological patterns.

All surgical procedures will be performed by the same surgeon, who was calibrated before the study and will be using the same surgical protocol for all participants. Before tooth extraction, participants from both groups will undergo local anaesthesia with mepivacaine 2%. A 15 mm periodontal probe will be used to measure from the inferior margin of an acrylic template to the bone crest at six different points: mesial, buccal, and distal (DB) (buccal region); and mesial, lingual, and distal (lingual region).All teeth will be extracted using a minimally traumatic procedure with no vertical releasing incisions. To avoid root and bony fractures, the molar teeth will be sectioned using a multilaminated drill. After exodontia, a rigorous inspection and curettage of the socket will be performed, followed by irrigation with sterile saline solution. The sockets of the test group will be filled with 1.2% SIM covered with polypropylene (PPP) membrane followed by cross suture to stabilize the membranes (n=15), while the sockets of the control group received the coverage with the PPP membrane (n=15). In both groups, the membrane will be intentionally exposed.

One week after extraction, an assessment of soft tissue healing around the sockets will be performed using the healing index system described by Landry et al. Furthermore, to assess postoperative pain the number of consumed analgesic tablets will be recorded, and a graphic rating scale will be filled and evaluated. In addition, after 90 days (T2), the patient will undergo a tomographic exam and the distances from the template to the crestal bone at six points will be measured before dental implant placement. Bone biopsy specimens obtained from representative cases will be process for qualitative and morphological analysis.

Data will be expressed as mean and 95% confidence interval. The Shapiro-Wilk or Kolmogorov-Smirnov normality test (alpha = 0.05) will be performed. The paired t test, analysis of variance (ANOVA), or Kruskal-Wallis test will be applied according to the number of groups. Tukey's or Dunn's multiple comparisons tests will be used to identify significant differences among the groups (p < 0.05). The Mann-Whitney unpaired test will be performed to analyse the effect of treatment on the healing index (p < 0.05). Nominal data will be evaluated by chi-square test.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged over 18 years
* Healthy patients with indication for dental extraction
* Teeth adjacent to the extraction site
* Patients willing to cooperate with the study and who have signed the informed consent form.

Exclusion Criteria:

* Patients showing periapical or periodontal infection
* Patients with severe systemic diseases
* Patients on medications such as chemotherapy, anticoagulants, corticosteroids, biphosphonates and immunosuppressant drugs,
* Patients who have chronic diseases decompensated (e.g. hypertension, diabetes, rheumatic diseases, renal, and hepatic)
* Patients with bone diseases, metabolic (osteomalacia, hypocalcemia and hypercalcemia).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2017-11-01 (Actual); Primary Completion 2020-03 (Estimated); Study Completion 2020-03 (Estimated)

PRIMARY OUTCOMES:
Dimensional change of the alveolar crest | 90 days
  Including soft and hard tissue, after clinical, histological and tomographic analysis

SECONDARY OUTCOMES:
Soft tissue healing | 1 week
  This analysis will be performed using the healing index system described by Landry et al.
Pain/discomfort | 1 week
  The number of consumed analgesic tablets will be recorded, and a graphic rating scale will be filled and evaluated

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Cruz, MSc, Principal Investigator — Fluminense Federal University
Locations (1):
- Dental Clinical Research Center of the Fluminense Federal University, Niterói, Rio de Janeiro, Brazil

REFERENCES:
- [Background] Landry R, Turnbull R, Howley T. Effectiveness of benzydamine HCL in the treatment of periodontal post-surgical patients. Res Clin Forums 10:105-118, 1998
- [Result] Moraschini V, Almeida DCF, Calasans-Maia JA, Diuana Calasans-Maia M. The ability of topical and systemic statins to increase osteogenesis around dental implants: a systematic review of histomorphometric outcomes in animal studies. Int J Oral Maxillofac Surg. 2018 Aug;47(8):1070-1078. doi: 10.1016/j.ijom.2017.12.009. Epub 2018 Jan 17. PMID 29352637
- [Result] Barone A, Ricci M, Tonelli P, Santini S, Covani U. Tissue changes of extraction sockets in humans: a comparison of spontaneous healing vs. ridge preservation with secondary soft tissue healing. Clin Oral Implants Res. 2013 Nov;24(11):1231-7. doi: 10.1111/j.1600-0501.2012.02535.x. Epub 2012 Jul 12. PMID 22784417
- [Result] Calasans-Maia M, Resende R, Fernandes G, Calasans-Maia J, Alves AT, Granjeiro JM. A randomized controlled clinical trial to evaluate a new xenograft for alveolar socket preservation. Clin Oral Implants Res. 2014 Oct;25(10):1125-30. doi: 10.1111/clr.12237. Epub 2013 Aug 13. PMID 23937306